CLINICAL TRIAL: NCT05142111
Title: Pilot Study on EEG and Behavioral Effects of Two Different Treatments on Sexual Life
Acronym: Seteb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Daniele Marinazzo, Scientific collaborator, IRCCS San Camillo, Venezia, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020.12
Record Dates: First submitted 2021-08-25; First posted 2021-12-02 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis; Spinal Cord Injuries
Keywords: sexuality
MeSH Terms: conditions — Multiple Sclerosis; Spinal Cord Injuries; Sexuality | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual therapy (Experimental): In the sessions a series of questions will be proposed to the subject, who will be free to answer or not, being able to express questions in turn. The sessions will last about 45 minutes, and will be held once a week, for a total of 6 sessions.
  Interventions: Behavioral: Therapy
- Mindfulness (Active Comparator): During the mindfulness treatment the subjects will be subjected to sessions in which they will be invited to relax, to become aware of the present moment, of their body, through exercises that involve breathing, attention, and visualization of the body.
  The sessions will last about 45 minutes, and will be held once a week, for a total of 6 sessions.
  Interventions: Behavioral: Therapy

INTERVENTIONS:
Behavioral: Therapy — Discussion with therapist

SUMMARY:
In this study patients with Multiple Sclerosis or Spinal Lesions will participate in two different types of treatments that aim to improve sexual and sentimental life. Behavioral (via questionnaires) and brain (via high-density electroencephalogram) effects associated with treatment will be studied.

DETAILED DESCRIPTION:
People with neurological diseases can experience sexual disorders that can affect their quality of life. There are cognitive treatments to improve these aspects, but their effectiveness is not clear. The aim of this study is to test the potential efficacy of two treatments (mindfulness and sezual therapy) in two neurological populations (patients with multiple sclerosis and patients with spinal injury). To verify the effects of the treatment, questionnaires and brain activity measurements, measured by electroencephalogram, will be used.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of MS or spinal injury.
* ability to sign informed consent.

Exclusion Criteria:

* other relevant previous neurological or psychiatric pathologies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of actual and perceived sexual health for females | Before and after treatment (circa 6 weeks)
  Assessed by means of a standardized questionnaire
  Female Sexual Dysfunction Questionnaire (Filocamo et al., 2014). 19 questions with 6 choices each. No maximum or minimum score defined. The experimenter evaluates the changes across sessions.
  This will be aggregated to other outcomes using factor analysis
Changes in quality of actual and perceived sexual health for males | Before and after treatment (circa 6 weeks)
  Assessed by means of a standardized questionnaire
  MSHQ- (The Male Sexual Health Questionnaire). Questionnaire on male sexual health (Ugolini, & Pescatori, 2005). 25 questions with 5 or 6 choices each. No maximum or minimum score defined. The experimenter evaluates the changes across sessions.
  This will be aggregated to other outcomes using factor analysis
Changes in erectile function | Before and after treatment (circa 6 weeks)
  Assessed by means of a standardized questionnaire
  IIEF5- (International Index of Erectile Function). Questionnaire aimed at calculating the International Index of Erectile Function (Rosen et al., 1997). 5 questions with scores 1 to 5. Outcome range 5-25. Lower scores indicate poorer outcomes.
  This will be aggregated to other outcomes using factor analysis
Changes in intimacy and sexuality | Before and after treatment (circa 6 weeks)
  Assessed by means of a standardized questionnaire
  MSISQ-15 (Multiple Sclerosis Intimacy and Sexuality Questionnaire). Questionnaire on Intimacy and Sexuality in People with a Medullary Injury (Monti et al., 2020). 15 items with scores 1 to 5 each. Outcome range 15-75. Higher scores indicate poorer outcomes.
  This will be aggregated to other outcomes using factor analysis

SECONDARY OUTCOMES:
Changes in brain spectral power after viewing neutral and erotic videos | Before and after treatment (circa 6 weeks)
  Changes in response of brain networks at rest and during viewing of emotional stimuli with sexual content. The recording will consist of 5 minutes of resting state (recording at rest). 8 total minutes of viewing of stimuli consisting of videos with an erotic and neutral emotional content. In particular, the subject will see two videos with an erotic content and two with an emotionally neutral content (the duration of each video is about 2 minutes). These stimuli will be selected from a standardized and validated visual battery for scientific studies presented in (Maffei & Angrilli, 2019).
  The spectral power across brain regions will be assessed by parametric spectral decomposition
  -presence and modulation of large scale patterns of correlated activity, assessed by means of measures of statistical dependency (correlation, mutual information)
Changes in Mutual Information between brain regions after viewing neutral and erotic videos | Before and after treatment (circa 6 weeks)
  Changes in response of brain networks at rest and during viewing of emotional stimuli with sexual content. The recording will consist of 5 minutes of resting state (recording at rest). 8 total minutes of viewing of stimuli consisting of videos with an erotic and neutral emotional content. In particular, the subject will see two videos with an erotic content and two with an emotionally neutral content (the duration of each video is about 2 minutes). These stimuli will be selected from a standardized and validated visual battery for scientific studies presented in (Maffei & Angrilli, 2019).
  The presence and modulation of large scale patterns of correlated activity, assessed by means of mutual information (minimal value zero, maximum value not univocally defined, depending on the data distribution), will be investigated.
Psychological Well-Being | Before and after treatment (circa 6 weeks)
  Assessed by means of a standardized questionnaire
  PWB (Psychological Well-Being Scale). Questionnaire aimed at defining the patient's psychological well-being profile through items that evaluate the dimensions of self-acceptance, autonomy, environmental control, life purpose, personal growth and positive relationships with others (Ruini et al., 2003). 42 items with scores 1-6 each. Outcome range 42-252. Higher values indicated better well-being.
  Questionnaire responses will be aggregated by factor analysis
Anxiety | Before and after treatment (circa 6 weeks)
  Assessed by means of a standardized questionnaire
  BAI (Beck Anxiety Inventory). Questionnaire consisting of 21 items that describe anxiety in its subjective, neurophysiological and autonomic aspects. (Sica & Ghisi, 2007; Starosta & Brenner, 2018). The BAI has also been found to be a tool with high sensitivity to anxiety levels in patients with multiple sclerosis (Watson et al., 2014). 21 items, with scores 1-4 each. Outcome range 21-84. Higher values indicate higher anxiety.
  Questionnaire responses will be aggregated by factor analysis
Changes in the assessment of the emotional response after viewing neutral and erotic videos | Before and after treatment (circa 6 weeks)
  Self-assessment questionnaires of the emotional content of stimuli, in particular the self-assessment manikin (SAM) will be used (Bradley MM, Lang PJ). With this questionnaire, through pictorial representations of "mannequins", the patient will be asked to evaluate his emotional reactions while watching the videos, in terms of the intensity of the emotions felt and the positive or negative values of the sensations experienced during the vision.
  9 mannequins for valence (score 1:sad, score 9: happy). 9 mannequins for arousal (increasing level 1 to 9).

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Marinazzo, PhD, Principal Investigator — Investigator
Locations (1):
- IRCCS San Camillo, Venice, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are trying to figure out compliance to EU GDPR, its interpretation in Italy, and the institutional requirements

REFERENCES:
- [Background] Chandler BJ, Brown S. Sex and relationship dysfunction in neurological disability. J Neurol Neurosurg Psychiatry. 1998 Dec;65(6):877-80. doi: 10.1136/jnnp.65.6.877. PMID 9854964
- [Background] Maffei A, Angrilli A. E-MOVIE - Experimental MOVies for Induction of Emotions in neuroscience: An innovative film database with normative data and sex differences. PLoS One. 2019 Oct 3;14(10):e0223124. doi: 10.1371/journal.pone.0223124. eCollection 2019. PMID 31581254
- [Background] McCabe MP. Evaluation of a cognitive behavior therapy program for people with sexual dysfunction. J Sex Marital Ther. 2001 May-Jun;27(3):259-71. doi: 10.1080/009262301750257119. PMID 11354931